CLINICAL TRIAL: NCT02288013
Title: Uterine Closure at C-section by Stratafix Tissue Control Device: Randomized Case-Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Zayed (Other)
Collaborators: Cairo University (Other); Johnson & Johnson Medical Companies (Industry)
Responsible Party: Sponsor-Investigator, Mohamed Zayed, Professor of Obstetrics and Gynecology Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IIS 13-207
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Cesarean Section
Keywords: Cesarean section; uterine closure technique; materials used

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratafix Tissue control device (Other): Closure of Uterine incision at C section
  Interventions: Procedure: Closure of uterine incision at C section
- Vicryl suture (Other): Closure of uterine incision at C section
  Interventions: Procedure: Closure of uterine incision at C section

INTERVENTIONS:
Procedure: Closure of uterine incision at C section — Closure of uterine incision at Cesarean section

SUMMARY:
Comparative study of the surgical outcome of 2-layers closure technique of uterine incision in Cesarean section using bidirectional barbed suture (Stratafix) and conventional suture material (Vicryl) regarding the time of closure and the need of secondary additional suturing or tearing of uterine muscles during suturing.

DETAILED DESCRIPTION:
A Randomized prospective case control study to evaluate the surgical outcome of using the new barbed bidirectional tissue controlling device in reducing the time and blood loss at uterine closure during C-Section. In addition, the need of additional sutures to control bleeding after the 2- layer closure is used and the occurrence of any tearing of the uterine muscles at the time closure of the uterine incision will be also studied. These will be the primary outcome measure and the secondary outcome measure will be factors related to the blood loss at the time of the uterine closure, surgical complications, duration of hospital stay, postoperative fever, and the number of sutures required to close the uterine incision.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant patients with an indication for delivery by C section

Exclusion Criteria:

* Patient refusing to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time needed to close the uterine incision | 6 minutes
  A model is set to evaluate success and failure according the ime needed to close the uterine incision if more or less than 6 minutes

SECONDARY OUTCOMES:
blood loss during uterine closure | intraoperative during uterine closure

OTHER OUTCOMES:
Duration of hospital stay | Six weeks following the cesarean delivery (completion of the postpartum period)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Z Ahmed, MD PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Cairo Governorate, Egypt